CLINICAL TRIAL: NCT05256316
Title: Risks of Bacterial and Fungal Superinfection in Patients With COVID-19 Stratified by New and Pre-existing Immunosuppression: a Retrospective, Observational, Multisite, Multinational Cohort Study
Brief Title: Risks of Bacterial and Fungal Superinfection in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Merck Sharp & Dhome (Australia) Pty. Ltd. (Unknown); Christian Medical College, Vellore, India (Other); Tan Tock Seng Hospital (Other); Royal Brisbane and Women's Hospital (Other Government); Siriraj Hospital (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/2021/QRBW/74171
Record Dates: First submitted 2022-02-24; First posted 2022-02-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: secondary infections; bacterial infections; fungal infections
MeSH Terms: conditions — COVID-19; Coinfection; Bacterial Infections; Mycoses | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Previously admitted COVID-19 patients in intensive care units: Infectious Diseases Physicians from participating hospitals will identify patients with COVID-19 admitted to their hospital who had an intensive care unit stay during the first 60 days after hospital admission.
  Interventions: Other: Previously admitted COVID-19 patients in intensive care units

INTERVENTIONS:
Other: Previously admitted COVID-19 patients in intensive care units — Exposure: this is a retrospective, observational study that does not include an intervention. Data collected for this study will be from previously hospitalized COVID-19 patients who had an intensive care unit stay during their admission

SUMMARY:
Infection with bacteria or fungi can be deadly. Often, these types of infections can lead to an increase in the severity of illness requiring intensive care unit (ICU) admission, prolonged duration of treatment and further risks associated with additional infections and superinfections. These are also called hospital acquired secondary infections. Patients who contract COVID-19 and require an ICU admission are at increased risk of contracting these secondary infections, and receive certain medications that can lower your body's immune response. In COVID-19 patients who require these treatments, it is unclear what affect these medications can have on developing an additional infection as well as the rate of recovery/survival. This study is evaluating the effect these medications have on the development of secondary infections and rate of survival of COVID-19 patients that have been admitted to ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission date from 1 July 2020 to 30 June 2021
* Positive test for COVID-19 collected within 1 week of admission date
* ICU admission within 60 days after hospital admission date

Exclusion Criteria:

* Hospital admission shorter than 5 days
* Persons younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously admitted COVID-19 patients admitted to Intensive Care Units
Sampling Method: Non-Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Describe the incidence, management and outcomes of secondary infections in COVID-19 patients admitted to intensive care units | Within the first 60 days of hospital admission
  Data collected from medical records of patients will include demographics, medical history, details of bacterial and fungal infections in the first 60 days after admission (includes aetiological pathogen, sample isolated from and antimicrobial susceptibility), treatment received for COVID-19 with antiviral or immunomodulatory therapy and disposition at 60 days from hospital admission
Compare clinical and microbiological outcomes based on treatment appropriateness in COVID-19 patients admitted to intensive care units | Within the first 60 days of hospital admission
  Data collected from medical records of patients will include demographics, medical history, details of bacterial and fungal infections in the first 60 days after admission (includes aetiological pathogen, sample isolated from and antimicrobial susceptibility), treatment received for COVID-19 with antiviral or immunomodulatory therapy and disposition at 60 days from hospital admission
Assess the use and effect of immune suppression in COVID-19 patients admitted to intensive care units. | Within the first 60 days of hospital admission
  Data collected from medical records of patients will include demographics, medical history, details of bacterial and fungal infections in the first 60 days after admission (includes aetiological pathogen, sample isolated from and antimicrobial susceptibility), treatment received for COVID-19 with antiviral or immunomodulatory therapy and disposition at 60 days from hospital admission

CONTACTS AND LOCATIONS:
Locations (5):
- University of North Carolina, Chapel Hill, North Carolina, United States
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia
- Christian Medical College, Vellore, India
- Tan Tock Seng Hospital, Singapore, Singapore
- Siriraj Hospital, Bangkok, Thailand